CLINICAL TRIAL: NCT06798714
Title: The Effect of Colchicine on the Occurrence of Atrial Fibrillation After Cardiac Surgery (CAFE)
Brief Title: The Effect of Colchicine on the Occurrence of Atrial Fibrillation After Cardiac Surgery
Acronym: CAFE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tomsk Cardiology Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Tomsk Cardiology Research Inst; Рег. № 123051500130-9: (Registry Identifier: DIAGNOSis AND TREATMENT OF CIRCULATORY SYSTEM DISEASES)
Record Dates: First submitted 2025-01-13; First posted 2025-01-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation; Coronary Artery Bypass Grafting; Colchicine
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation | interventions — Anti-Inflammatory Agents, Non-Steroidal; Colchicine

STUDY DESIGN:
Intervention Model Description: Group 1 (n=70): Patients who underwent pericardial fenestration during CABG surgery and received perioperative colchicine.
  Group 2 (n=70). Patients operated on using the standard technique (CABG without pericardial fenestration) and receiving NSAIDs in the postoperative period.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Standard technique without performing the pericardial fenestration procedure intraoperatively. Standard postoperative treatment
  Interventions: Drug: NSAID
- Experimental group (Experimental): Pericardial fenestration during coronary artery bypass grafting using the original technique.
  Colchicine (Colchicum-dispert) administration 4 hours before surgery and for 10 days after surgery
  Interventions: Drug: Colchicine 0.5 MG

INTERVENTIONS:
Drug: NSAID — standard CABG without performing pericardial fenestration intraoperatively
  Other Names: non-steroidal anti-inflammatory drugs
  Arms: Control group
Drug: Colchicine 0.5 MG — Colchicine will be prescribed in a dose of 500 micrograms 4 hours before surgery and 500 micrograms 2 times a day for 10 days after surgery with pericardial fenestration
  Other Names: Colchicum-dispert
  Arms: Experimental group

SUMMARY:
Development of a new comprehensive method for perioperative prevention of atrial fibrillation paroxysms in cardiac surgery patients at the hospital stage.

It is planned to recruit 70 patients who will undergo pericardial fenestration during the operation using the original technique during coronary artery bypass grafting (Patent No. 2647626 C1 Russian Federation), and will be prescribed colchicine (the drug "Colchicum-dispert") in the perioperative period in order to prevent the development of paroxysms of atrial fibrillation in the postoperative period, and 70 cardiac surgery patients operated on using the standard technique (without performing the pericardial fenestration procedure intraoperatively), receiving non-steroidal anti-inflammatory drugs in the postoperative period.

DETAILED DESCRIPTION:
Study type: observational, analytical, cohort, prospective. Purpose: development of a new comprehensive method for perioperative prevention of atrial fibrillation paroxysms in cardiac surgery patients at the hospital stage.

Objectives:

1. To assess the risk factors that influence the development of atrial fibrillation in the early postoperative period;
2. To conduct a comparative analysis of various therapy methods to reduce the risk of developing atrial fibrillation paroxysms in the early postoperative period in cardiac surgery patients.

To solve the set tasks, it is planned to conduct a cohort prospective observational study of patients with coronary artery disease who underwent coronary artery bypass grafting with cardiopulmonary bypass.

Duration of the study - 1,5 years. The observation period for patients is the hospital postoperative period after CABG.

The study is planned to include 140 patients diagnosed with coronary heart disease. The diagnosis will be established on the basis of medical records and coronary angiography. Indications for CABG surgery will be determined by a consulting cardiac surgeon in accordance with the current Clinical Guidelines of the Ministry of Health of the Russian Federation "Stable ischemic heart disease" (2020).

Patients should be over 18 years old. It is planned to recruit 70 patients who will undergo pericardial fenestration during coronary artery bypass grafting using the original technique (Patent No. 2647626 C1 Russian Federation), and will be prescribed colchicine (the drug "Colchicum-dispert") in the perioperative period in order to prevent the development of paroxysms of atrial fibrillation in the postoperative period, and 70 cardiac surgery patients operated on using the standard technique (without performing the pericardial fenestration procedure intraoperatively), receiving non-steroidal anti-inflammatory drugs in the postoperative period. Diclofenac will be used as an NSAID in the postoperative period at a daily dose of 100 mg (orally). Colchicine (trade name of the drug "Colchicum-dispert") will be prescribed in a dose of 500 micrograms 4 hours before surgery and 500 micrograms 2 times a day for 10 days after surgery. Since the drug is not registered for the prevention of atrial fibrillation in the postoperative period, its prescription will be decided by a council of doctors, including at least 3 people (head of the department, attending physician, and research physician).

Safety evaluation Since no medical studies or interventions will be carried out in addition to what the patient should receive during standard examination and treatment, participation in this study does not entail any risks and threats to the patient.

The safety endpoints of standard treatment for this disease will be analyzed. Statistical analysis Statistical analysis of data will be carried out in the STATISTICA 10 StatSoft program. Inc. 1984-2011 (USA). Quantitative values will be displayed as median and quartiles Me [25;75]. Comparison of quantitative characteristics between groups will be performed using the Mann-Whitney U-test. Fisher's exact test will be used to compare qualitative characteristics. Differences will be considered statistically significant at p < 0.05.

Ethical and legal issues of the study:

The study was approved by the Biomedical Ethics Committee at Cardiology Research Institute of Tomsk National Research Medical Center.

All patients must sign an informed consent form allowing the use of information about their examination and treatment for scientific purposes with subsequent publication of materials in the open press. The study will be conducted in accordance with the current version of the Declaration of Helsinki, the provisions of the National Standard of the Russian Federation GOST R52379-2005 on Good Clinical Practice dated April 1, 2006, the Order of the Ministry of Health of the Russian Federation dated April 1, 2016 No. 200n "On approval of the rules of good clinical practice" and the provisions of Good Clinical Practice (GCP).

The procedure for informing study subjects and obtaining written consent from them will be carried out in accordance with GCP standards.

ELIGIBILITY:
Inclusion Criteria:

1. Elective coronary artery bypass grafting on pump;
2. signed informed consent to participate in the study.

Exclusion Criteria:

1. Reduced left ventricular ejection fraction (≤35%);
2. Valvular heart disease requiring surgical correction;
3. Liver failure with an increase in liver transaminases ≥1.5 times;
4. Renal failure (GFR<35 mL/min/1.73 m2 calculated with CKD-EPI);
5. Permanent, persistent or paroxysmal atrial fibrillation;
6. Previously implanted pacemaker;
7. Hypersensitivity to colchicine;
8. Neutropenia;
9. History of alcoholism;
10. Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of atrial fibrillation paroxysms (percent) | From the date of randomization until the date of discharge from hospital (from 10 days to 4 weeks)
  Differences between groups in the incidence of atrial fibrillation paroxysm development (percent)

SECONDARY OUTCOMES:
Incidence of pneumonia (percent) | From the date of randomization until the date of discharge from hospital (from 10 days to 4 weeks)
  Differences between groups in the incidence of pneumonia development (percent)
Incidence of mediastinitis (percent) | From the date of randomization until the date of discharge from hospital (from 10 days to 4 weeks)
  Differences between groups in the incidence of mediastinitis development (percent)
Level of C-reactive protein (CRP) (mg/L) | 10 days
  The difference in the levels of C-reactive protein (CRP) (mg/L) between the study groups after surgery
Level of aspartate aminotransferase (AST) (U/L) | 10 days
  The difference in the levels of The difference in the levels of aspartate aminotransferase (AST) (U/L) between the study groups after surgery
Level of alanine aminotransferase (ALT) (U/L) | 10 days
  The difference in the levels of The difference in the levels of alanine aminotransferase (ALT) (U/L) between the study groups after surgery
Level of blood creatinine (µmol/L) | 10 days
  The difference in the levels of blood creatinine (µmol/L) between the study groups after surgery
Pericardial fluid volume (mL) | 10 days
  The difference in the volume of pericardial fluid (mL) between the study groups after surgery
Pleural fluid volume (mL) | 10 days
  The difference in the volume of pleural fluid (mL) between the study groups after surgery
Incidence of gastrointestinal disorders (percent) | 10 days
  Differences between groups in the incidence of nausea and/or diarrhea after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Y Vechersky, PhD, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Center, Russian Academy of Sciences, Tomsk, Russia, Tomsk, Russia

REFERENCES:
- [Derived] Diakova ML, Kuznetsov MS, Vechersky YY, Kim EB, Zyryanov SV, Petlin KA, Kozlov BN. A Combined Approach to the Prevention of Postoperative Atrial Fibrillation in Cardiac Surgery. Biomedicines. 2025 Aug 17;13(8):1999. doi: 10.3390/biomedicines13081999. PMID 40868251